CLINICAL TRIAL: NCT00728039
Title: Quality of Life, Coping and Psychological Symptoms in Children and Adolescents With Cyclic Vomiting Syndrome
Brief Title: Quality of Life (QOL), Coping and Psychological Symptoms in Children and Adolescents With Cyclic Vomiting Syndrome
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, B Li, Associate Professor, Medical College of Wisconsin
Other Study IDs: 07/82; GC 399
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Vomiting Syndrome
Keywords: Youth; Consensus; Criteria; CVS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
1. Characterize the quality of life of young children with CVS (i.e., psychological, social, physical, school functioning) and the impact of the child's illness on the parent's and family's quality of life (i.e., emotional, social, cognitive functioning, communication, worry, daily activities and family relationships).
2. Assess symptoms of depression, anxiety, ADHD and behavioral problems in what our preliminary data suggests is a psychiatrically vulnerable population.
3. Evaluate the associations between quality of life and psychiatric symptoms and the frequency and intensity of CVS attacks.
4. Use the data generated from this study to develop a psychosocial intervention targeted at young children with CVS and their families who evidence risk for functional disability, with the aim of intervening as early as possible to limit the psychological and social morbidity experienced by children with CVS and their and families.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CVS

Exclusion Criteria:

* Children and parents who are not English speaking
* Youth with significant developmental delay, mental retardation, psychotic symptoms, or other significant mental impairments and those with other major medical disorders such as IDDM, congenital heart disease, cystic fibrosis, etc.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 9-10 will complete 5 questionnaires Adolescents aged 11-18 will complete 6 questionnaires Youth aged 11-18 will fill out an additional questionnaire that asks how they cope with stress related to CVS symptoms Parents will complete 4 questionnaires
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2007-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Characterize the quality of life of youth with CVS as well as the strategies they use to cope with stress, their strengths and vulnerabilities, and to assess symptoms of depression and anxiety in these at risk youth. | Two years

SECONDARY OUTCOMES:
Evaluate the associations among coping strategies the frequency and intensity of CVS attacks to determine if particular coping styles and personal characteristics are associated illness severity, psychiatric co-morbidity and quality of life. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Sally E Tarbell, PhD, Principal Investigator — Medical College of Wiconsin